CLINICAL TRIAL: NCT01879033
Title: Effect Of Obesity And Hyperglycemia on Endothelial Function in Inner City Bronx Adolescents
Brief Title: Endothelial Function in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-07-219E
Record Dates: First submitted 2013-06-05; First posted 2013-06-17 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Insulin Resistance; Glucose Intolerance; Obesity; Atherosclerosis
Keywords: Obesity; endothelial function; Rh-PAT; adipocytokines
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Obesity; Atherosclerosis | interventions — Glucose; Insulin; Lipids; Adipokines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese adolescents (Active Comparator): Those with BMI more than or equal to 95th percentile. This group was further divided into two subgroups on the basis of Oral Glucose Tolerance Test (OGTT) into normal and impaired glucose tolerance groups. Reactive hyperemia peripheral artery tonometry (Rh-PAT)score and blood levels for glucose, insulin, lipids and adipocytokines will be measured in the study.
  Interventions: Other: Reactive hyperemia peripheral artery tonometry (Rh-PAT); Other: Blood levels for glucose, insulin, lipids and adipocytokines
- Lean adolescents (Placebo Comparator): BMI between 5th-85th percentile.Reactive hyperemia peripheral artery tonometry (Rh-PAT)score and blood levels of glucose, insulin, lipids and adipocytokines will be measured in the study.
  Interventions: Other: Reactive hyperemia peripheral artery tonometry (Rh-PAT); Other: Blood levels for glucose, insulin, lipids and adipocytokines

INTERVENTIONS:
Other: Reactive hyperemia peripheral artery tonometry (Rh-PAT) — Pulse volume is measured by a finger plethysmographic device which are sensed by a pressure transducer and transferred to a computer where the signal is amplified, displayed and stored (EndoPAT, Itamar Medical). Fingertip probes are placed on the index finger of both hands and 5 minutes of baseline recording are obtained. Blood flow is then occluded in one arm for 5 minutes, using a standard blood pressure cuff. Recording continues in both fingers during occlusion and for 5 minutes after release of the cuff. The RH-PAT index is calculated as the ratio of the average pulse amplitude in the post-hyperemic phase divided by the average baseline amplitude, with normalization to the signal in the control arm to compensate for any systemic changes.
  Other Names: Endopat
Other: Blood levels for glucose, insulin, lipids and adipocytokines — A fasting laboratory evaluation will include chemistry panel (basic metabolic, liver function tests), CBC, lipid profile, urinalysis and HbA1c. All obese recruited subjects after a 12 hour fast will undergo an OGTT using a glucose load of 1.75 g/kg body weight with a maximum of 75 g. Blood samples will be collected for insulin, glucose, leptin, adiponectin, hsCRP and FFA. Serum and urine will be stored at -70 degrees Centigrade for measuring markers of oxidative stress and adipocytokines (including TNF-α, PAI-1)

SUMMARY:
Childhood obesity is perhaps the most significant public health problem in the most developed countries and is rapidly becoming so in developing countries. National Health and Nutrition Examination Survey data shows a 3-fold increase in the prevalence of obesity in childhood, over past few decades. Furthermore, childhood obesity has markedly contributed to the prevalence of the metabolic syndrome and type 2 diabetes in U.S. children. Alarmingly, there is increasing evidence that atherosclerosis develops silently during childhood in obese children. In the Bogalusa Heart Study, pediatric autopsy studies showed a clear relationship between the number and severity of risk factors, principally obesity, with atherosclerosis in both the aorta and coronary arteries. Increased intimal medial thickness (IMT) was not present among obese adults who had been normal weight as children, emphasizing the cumulative effects of childhood obesity persisting into adulthood. Thus, the need for primary prevention of cardiovascular disease beginning in childhood is strongly suggested.

DETAILED DESCRIPTION:
Following informed consent, a detailed history and physical examination will be performed including supine blood pressure taken twice after a 20 minute period of rest, height (using Harpenden stadiometer) to the nearest 0.1 cm and weight will be measured to the nearest 0.1 kg with a balance scale, pubertal staging using the method of Marshall and Tanner, waist measurement obtained at the minimal circumference of the abdomen, hip measurements with a plastic tape while the subject is standing and recorded at the widest diameter over the greater trochanters. BMI (kg/m2) and waist to hip ratio will be calculated. Screening labs in all recruited subjects: A fasting laboratory evaluation will include chemistry panel (basic metabolic, liver function tests), Complete Blood Count (CBC), lipid profile, urinalysis and HbA1c. All obese recruited subjects after a 12 hour fast will undergo an OGTT using a glucose load of 1.75 g/kg body weight with a maximum of 75 g. Blood samples will be collected for insulin, glucose, leptin, adiponectin, High sensitive C-reactive protein (hsCRP) and Free Fatty Acids (FFA). Serum and urine will be stored at -70 (degree Centigrade)C for measuring markers of oxidative stress and adipocytokines (including Tumor Necrosis Factor (TNF)-α, Plasminogen Acivator Inhibitor (PAI)-1) for future studies depending on the funding availability.

Subjects who fulfill the study criteria would be admitted to Clinical Research Center to evaluate endothelial function by RH-PAT.

RH-PAT for endothelial function Reactive hyperemia peripheral arterial tonometry (RH-PAT) is a noninvasive technique used to assess peripheral microvascular endothelial function by measuring changes in digital pulse volume during reactive hyperemia (Bonetti, Kuvin). Pulse volume is measured by a finger plethysmographic device that allows isolated detection of pulsatile arterial volume changes, which are sensed by a pressure transducer and transferred to a computer where the signal is amplified, displayed and stored (EndoPAT, Itamar Medical). Studies are performed with the patient at rest, in a comfortable, thermo neutral environment. Fingertip probes are placed on the index finger of both hands and 5 minutes of baseline recording are obtained. Blood flow is then occluded in one arm for 5 minutes, using a standard blood pressure cuff. Recording continues in both fingers during occlusion and for 5 minutes after release of the cuff. The RH-PAT index is calculated as the ratio of the average pulse amplitude in the post-hyperemic phase divided by the average baseline amplitude, with normalization to the signal in the control arm to compensate for any systemic changes.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age range of 12-18 years
* For the lean group, age and sex matched subjects with BMI between 5th-85th percentiles
* Obese group defined as BMI ≥95th percentile. These will further be subgrouped into those with normal and those with abnormal glucose tolerance normal glucose tolerance (NGT) defined as fasting glucose level<100mg/dl and a 2 hour postprandial glucose level<140mg/d and abnormal OGTT defined as fasting level ≥100mg/dl and/or 2hr ≥140 using a glucose load of 1.75 g/kg body weight (max 75 g).Hence, we will

Exclusion Criteria:

-

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
RH-Pat score | 2 weeks after Screening Visit
  After Screening visit, the subjects were assessed for endothelial function using Rh-PAT.

SECONDARY OUTCOMES:
insulin levels | Visit 1 (two(2) weeks after Screening Visit)
  Subjects were assesses for insulin level on Visit 1. Lean subjects only had fasting levels of insulin, while obese had 2 hour Oral glucose tolerance test.
Lipid Profile | Visit 1 (two(2) weeks after Screening Visit)
  Subjects were assessed for fasting cholesterol, Low density lipoprotein (LDL), High density lipoprotein (HDL) and Triglyceride levels during the visit 1.
Adipocytokine levels | Visit 1 (two(2) weeks after Screening Visit)
  Subjects were assessed for levels of adipocytokines which include Leptin, Adiponectin, Tumor Necrosis Factor (TNF)- alfa, Interleukin (IL)-6 during the Visit 1.
Glucose levels | Visit 1 (two(2) weeks after Screening Visit)
  Subjects were assesses for glucose levels on Visit 1. Lean subjects only had fasting levels of glucose, while obese had 2 hour Oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Chhavi Agarwal, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Albert Einstein College of Medicine West Campus Clinical Research Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Agarwal C, Cohen HW, Muzumdar RH, Heptulla RA, Renukuntla VS, Crandall J. Obesity, hyperglycemia and endothelial function in inner city Bronx adolescents: a cross-sectional study. Int J Pediatr Endocrinol. 2013 Oct 29;2013(1):18. doi: 10.1186/1687-9856-2013-18. PMID 24164965